CLINICAL TRIAL: NCT02864836
Title: Study of the ISotopic Repartition of cOpper in Head and Neck TumOral and lymPhomatous pathologiEs
Brief Title: Study of Copper Isotope in Head and Neck Cancer
Acronym: ISOTOPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: Ecole Normale Supérieure de Lyon (Unknown)
Responsible Party: Sponsor
Other Study IDs: RT-14
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Tumors
Keywords: Copper; isotopic distribution; cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Urine Saliva cancer tissue healthy tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with head or neck cancer: Samples collection
  Interventions: Procedure: Samples collection
- Patients with lymphoma: Samples collection
  Interventions: Procedure: Samples collection
- Patients without tumoral pathology: Samples collection
  Interventions: Procedure: Samples collection

INTERVENTIONS:
Procedure: Samples collection — 5 samples collected for each patient (tumor biopsy, healthy tissue around the tumor, blood, urine and saliva), quantification of isotopes, measure of mRNA expression of proteins 4 samples for each patient (healthy tissue, blood, urine and saliva), quantification of isotopes, measure of mRNA expression of proteins

SUMMARY:
The distribution of stable (non-radioactive) isotopes in living organisms is increasingly studied, in particular the zinc (Zn), copper (Cu) and iron (Fe), not only in primitive organisms, but also in mammals.

The scientific community shows a growing interest in the study of the isotopic distribution of Cu in humans: this distribution can vary according to gender or nutrition. Concerning pathology, the isotopic distribution of Cu seems interesting in Wilson's disease or in cirrhosis.

Additionally, a promising area of study focuses on the role of Cu in cancerous tumors, neoangiogenesis, the mechanisms of free radicals reduction and signaling pathways.

Head and neck cancers are sensitive to platinum salts. Links between platinum and Cu are important: platinum penetrates into the cell through a Cu receptor, it interacts with the regulation mechanisms of Cu and platinum.

Preliminary studies suggest a variation of the measurable isotopic distribution of Zn in patients with breast tumor and of Cu in patients presenting breast as well as colorectal tumors.

The Larner et al. study suggest a promising role of Zn in breast cancer, indeed, results highlight a variation of distribution of Zn in 10 breast tumors. Concerning the study of Télouk et al. on 8 patients presenting colorectal tumors and 20 patients presenting breast tumors, results are in favor of an increase of mortality when Cu 65 is decreased in the serum and the isotopic modifications happen earlier than usual modifications of biochemical tumor markers such as: carbohydrate antigen (CA) 19.9, Carcinoma Antigen (CA) 15.3, Carcinoembryonic antigen (CEA).

Currently, there is no information about the distribution of the stable isotopes of Cu in head and neck tumors.

The objective of the study is to determine if the distribution of 65Cu / 63Cu is modified in tumoral tissues compared to healthy tissues. The isotopic distribution of the Cu in 2 tumor types, head and neck tumors and lymphomas, will be also investigated in order to determine if this distribution is specific of a tumor type or not.

In case of positivity of this variation, the prognostic interest of these parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of head and neck malignant tumors or clinical diagnosis of head and neck lymphoma requiring sampling for diagnosis or clinical diagnosis of a non tumoral ENT pathology requiring surgery

Exclusion Criteria:

Refusal of consent

Inability to consent

Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups of patients will be involved in this study:
  * Patients with head and neck malignant tumors,
  * Patients with lymphoma,
  * Patients without tumoral ENT pathology
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Ratio of the different stable isotopes of copper in the various samples and groups | Baseline

SECONDARY OUTCOMES:
Patient survival rate | at 5 years
mRNA expression level of proteins involved in copper metabolism assessed by Polymerase chain reaction (PCR) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bartaire, PhD, Principal Investigator — GHICL
Locations (2):
- France (2):
  - GHICL, Lille
  - ENS Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No